CLINICAL TRIAL: NCT01701934
Title: Impact of Roflumilast on Visceral Adiposity and MetaBolic Profile in Chronic Obstructive Lung Disease: a Randomized and Controlled Trial: the RAMBO Trial.
Brief Title: Impact of Roflumilast on Visceral Adiposity and Metabolic Profile in Chronic Obstructive Pulmonary Disease
Acronym: RAMBO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The recruitment of the study was prematurely stopped in July 2014 for the following reason; no more study medication.
Sponsor: Laval University (Other)
Collaborators: Innovair (Unknown); Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RAMBO
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Metabolic Syndrome
Keywords: COPD; Intrabdominal adiposity; Body composition; Triglycerides; Cholesterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Metabolic Syndrome | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Roflumilast (Experimental): Roflumilast 500 mcg, once daily for 6 months
  Interventions: Drug: Roflumilast
- Placebo pill (Placebo Comparator): Placebo pill, once daily for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — 500 mcg, oral, once daily for 6 months
  Other Names: DAXAS
  Arms: Roflumilast
Drug: Placebo — One placebo pill daily, for 6 months
  Other Names: Inactive comparator
  Arms: Placebo pill

SUMMARY:
The purpose of this study is to determine whether roflumilast can improve metabolic profile and reduce visceral adiposity in patients with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Although underweight has been the traditional nutritional concern in patients with COPD, overweight and obesity are becoming important issues in this disease. In a rehabilitation study, investigators found that 66% of patients with moderate to severe COPD were either overweight or obese according to the WHO obesity classification (BMI ≥ 25 kg/m2). Obesity and COPD being two frequent conditions, it is important to understand the nature of their interactions.

Obesity, particularly in its visceral form is associated with a plethora of metabolic consequences that increases the risk of cardiovascular diseases. This would seem relevant to COPD which is in itself an important risk factor for cardiovascular diseases. The presence of obesity, particularly visceral obesity, may thus define in patients with COPD a clinical phenotype at high risk of cardiovascular diseases. In this context, it is relevant to note that the prevalence of metabolic syndrome is increased in COPD. Although fat distribution has not been precisely assessed in COPD studies, increased waist circumference is common in this disease suggesting that visceral obesity is part of the obesity syndrome seen in COPD.

Given the relationship between COPD, obesity and the metabolic syndrome and cardiovascular diseases, it is tempting to suggest that visceral obesity is likely to be frequent in COPD (as in the general population) and that the profound metabolic and inflammatory perturbations associated with this form of overweight/obesity could play a central role in the link between COPD and cardiovascular diseases.

Roflumilast, a Phosphodiesterase-4 inhibitor, has been recently evaluated as an anti-inflammatory medication in patients with COPD. Roflumilast, alone or in combination with long-acting bronchodilators, provide modest but significant improvement in lung function along with reductions in the rate of exacerbation in patients with moderate to severe COPD. A very interesting observation that was made in these 12-month duration studies was that the use of roflumilast was associated with an average reduction in body weight of 2 kg that took place during the first 6 months of the trials and remained relatively stable throughout the rest of the trials. The mechanisms and the precise effects of roflumilast on body composition and adipose tissue distribution have not been studied in great detail. However, available data suggest that roflumilast induces a preferential loss in body fat mass in comparison to fat-free mass. It remains to be seen whether roflumilast specifically affects visceral versus subcutaneous adipose tissue. The improved insulin sensitivity reported in one study in the presence of an apparently trivial weight loss (0.7 kg compared to placebo) may suggest that a selective loss of visceral adipose tissue may have been produced in response to roflumilast therapy.

These observations, although not definitive, suggest that roflumilast could be used not only to treat the respiratory component of COPD but also to modulate the metabolic aspect of this disease including visceral adiposity, features of the metabolic syndrome and significant co-morbidities of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Gave an informed consent
* Forced expiratory volume in 1 second < 80% predicted
* Forced expiratory volume in 1 second / Forced vital capacity < 70%
* No exacerbation in the last 4 weeks
* Current or ex-smoker
* Smoking history of at least 10 pack/year
* Body mass index of at least 25 kg/m2
* Waist circumference of at least 94 cm
* Fasting blood triglycerides of at least 1.7 mmol/L

Exclusion Criteria:

* Any significant pulmonary pathology other than COPD
* Under oxygen therapy more than 12 hours per day
* More than 2 exacerbation episodes in the last 12 months
* The patient is currently participating to the active phase of a rehabilitation program
* Patient has been under roflumilast therapy prior to enrollment
* Unstable hypertriglyceridemia or hypercholesterolemia
* Under diabetes therapy (hypoglycemic agent or insulin)
* Cancer history in the last 5 years (except basal cell carcinoma)
* Moderate or severe hepatic impairment
* Used prednisone or systemic corticosteroids in the last 4 weeks

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-02; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change in intrabdominal adiposity | At baseline and 6 months later
  Measured by CT scan.

SECONDARY OUTCOMES:
Change in body mass index | At baseline and 6 months later
Change in waist circumference | At baseline and 6 months later
Change in waist-to-hip circumference ratio | At baseline and 6 months later
Change in blood metabolic profile | At baseline and 6 months later
  Blood glucose, insulin, triglycerides, apolipoprotein B, LDL/HDL cholesterol, C-reactive protein will be measured.
Change in body composition | At baseline and 6 months later
  As measured by dual-energy X-ray absorptiometry (DEXA).
Change in subcutaneous adiposity | At baseline and 6 months later
  As measured by CT scan.
Change in liver fat | At baseline and 6 months later
  As measured by CT scan

CONTACTS AND LOCATIONS:
Overall Officials: François Maltais, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (5):
- Canada (5):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Montreal Chest Institute, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec
  - Hôpital régional de Saint-Jérôme, Saint-Jérôme, Quebec

REFERENCES:
- [Background] Sava F, Laviolette L, Bernard S, Breton MJ, Bourbeau J, Maltais F. The impact of obesity on walking and cycling performance and response to pulmonary rehabilitation in COPD. BMC Pulm Med. 2010 Nov 6;10:55. doi: 10.1186/1471-2466-10-55. PMID 21054892
- [Background] Despres JP, Lemieux I. Abdominal obesity and metabolic syndrome. Nature. 2006 Dec 14;444(7121):881-7. doi: 10.1038/nature05488. PMID 17167477
- [Background] Sin DD, Man SF. Why are patients with chronic obstructive pulmonary disease at increased risk of cardiovascular diseases? The potential role of systemic inflammation in chronic obstructive pulmonary disease. Circulation. 2003 Mar 25;107(11):1514-9. doi: 10.1161/01.cir.0000056767.69054.b3. PMID 12654609
- [Background] Marquis K, Maltais F, Duguay V, Bezeau AM, LeBlanc P, Jobin J, Poirier P. The metabolic syndrome in patients with chronic obstructive pulmonary disease. J Cardiopulm Rehabil. 2005 Jul-Aug;25(4):226-32; discussion 233-4. doi: 10.1097/00008483-200507000-00010. PMID 16056071
- [Background] Lam KB, Jordan RE, Jiang CQ, Thomas GN, Miller MR, Zhang WS, Lam TH, Cheng KK, Adab P. Airflow obstruction and metabolic syndrome: the Guangzhou Biobank Cohort Study. Eur Respir J. 2010 Feb;35(2):317-23. doi: 10.1183/09031936.00024709. Epub 2009 Jul 2. PMID 19574332
- [Background] Fabbri LM, Calverley PM, Izquierdo-Alonso JL, Bundschuh DS, Brose M, Martinez FJ, Rabe KF; M2-127 and M2-128 study groups. Roflumilast in moderate-to-severe chronic obstructive pulmonary disease treated with longacting bronchodilators: two randomised clinical trials. Lancet. 2009 Aug 29;374(9691):695-703. doi: 10.1016/S0140-6736(09)61252-6. PMID 19716961
- [Background] Calverley PM, Rabe KF, Goehring UM, Kristiansen S, Fabbri LM, Martinez FJ; M2-124 and M2-125 study groups. Roflumilast in symptomatic chronic obstructive pulmonary disease: two randomised clinical trials. Lancet. 2009 Aug 29;374(9691):685-94. doi: 10.1016/S0140-6736(09)61255-1. PMID 19716960